CLINICAL TRIAL: NCT02086045
Title: A NON-RANDOMIZED, CONSECUTIVE ENROLLMENT EVALUATION OF THE DESolve® NOVOLIMUS ELUTING BIORESORBABLE CORONARY SCAFFOLD SYSTEM IN THE TREATMENT OF PATIENTS WITH DE NOVO NATIVE CORONARY ARTERY LESIONS
Brief Title: Elixir Medical Clinical Evaluation of the DESolve® Novolimus Eluting Bioresorbable Coronary Scaffold System - The DESolve Nx Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1003
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DESolve Novolimus Eluting Bioresorbable Coronary Scaffold (Other): DESolve Scaffold
  Interventions: Device: DESolve Novolimus Eluting Bioresorbable Coronary Scaffold System

INTERVENTIONS:
Device: DESolve Novolimus Eluting Bioresorbable Coronary Scaffold System — percutaneous coronary

SUMMARY:
To evaluate the safety, performance and efficacy of the Elixir DESolve® Novolimus Eluting Bioresorbable Coronary Scaffold System (BCSS) in patients with a single de novo native coronary artery lesion designated the target lesion and up to one non-target lesion located in a separate epicardial vessel.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age and for the 35-patient subset, patients must be over the age of 50
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the DESolve Nx Novolimus Eluting BCSS and he/she provides written informed consent, as approved by the appropriate Ethics Committee of the respective clinical site, prior to any clinical study related procedure
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or electrocardiogram (ECG) changes consistent with ischemia)
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
* Patient must agree to undergo all clinical study required follow-up visits, angiograms, and as applicable, IVUS, OCT, MSCT and coronary vasomotion testing
* Patient must agree not to participate in any other clinical study for a period of two years following the index procedure

Angiographic Inclusion Criteria:

Target lesion must be located in a native coronary artery with a nominal vessel diameter of between 2.75 and 3.5 mm assessed by online QCA

* Target lesion must measure ≤ 14 mm in length
* Target lesion must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 90% with a TIMI flow of ≥ 1
* Percutaneous intervention of lesions in the target vessel if:

  1. Not part of a clinical investigation
  2. ≥ 6 months prior to the study index procedure
  3. ≥ 9 months after the study index procedure (planned)
  4. Previous intervention was distal to and >10mm from the target lesion

Exclusion Criteria:

* Patient has a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure and CK and CK-MB have not returned within normal limits at the time of procedure
* Patient is currently experiencing clinical symptoms consistent with AMI
* Patient requires the use of any rotablator intervention during the index procedure
* Patient has current unstable arrhythmias
* Patient has a known left ventricular ejection fraction (LVEF) < 30%
* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
* Patient is receiving chronic anticoagulation therapy (e.g., heparin, coumadin) that cannot be stopped and restarted according to local hospital standard procedures.
* Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, Novolimus, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease.
* Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, or patient on dialysis)
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
* Patient is already participating in another clinical study
* Women of childbearing potential who have not undergone surgical sterilization or are not post-menopausal (defined as amenorrheic for at least one year) as well as women who are pregnant or nursing
* Patient is unable to give their consent, is legally incompetent, or is institutionalized by virtue of an order issued by the courts or other authority

Angiographic Exclusion Criteria

* Target lesion(s) meets any of the following criteria:

  1. Aorto-ostial location
  2. Left main location
  3. Located within 5 mm of the origin of the LAD or LCX
  4. Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
  5. Lesion involving a side branch >2mm in diameter or bifurcation
  6. Previous placement of a scaffold proximal to or within 10 mm of the target lesion
  7. Total occlusion (TIMI flow 0), or TIMI flow < 1
  8. Excessive tortuosity proximal to or within the lesion
  9. Angulation (≥ 45o) proximal to or within the lesion
  10. Calcification moderate or heavy
  11. Previous intervention restenosis
* The target vessel contains visible thrombus
* Another clinically significant lesion (>40%) is located in the same major epicardial vessel as the target lesion
* Patient has a high probability that a procedure other than pre-dilatation and scaffolding and (if necessary) post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon or brachytherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Clinically-indicated major adverse cardiac events (MACE) | 6 months
  cardiac death, target vessel MI, clinically indicated TLR
Late Lumen Loss | 6 month
  MLD post procedure - MLD at follow-up

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 1 month
  cardiac death, target vessel MI, clinically indicated TLR
Major Adverse Cardiac Events | 12 months
  cardiac death, target vessel MI, clinically indicated TLR
Major Adverse Cardiac Events | 24 months
  cardiac death, target vessel MI, clinically indicated TLR
Major Adverse Cardiac Events | 3 years
  cardiac death, target vessel MI, clinically indicated TLR
Major Adverse Cardiac Events | 4 years
  cardiac death, target vessel MI, clinically indicated TLR
Major Adverse Cardiac Events | 5 months
  cardiac death, target vessel MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 1 month
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 6 months
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 1 year
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 2 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 3 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 4 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Lesion Failure (TLF) | 5 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Vessel Failure (TVF) | 1 year
  cardiac death, MI, clinically indicated TVR
Clinically-Indicated Target Vessel Failure (TVF) | 2 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Vessel Failure (TVF) | 3 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Vessel Failure (TVF) | 4 years
  cardiac death, MI, clinically indicated TLR
Clinically-Indicated Target Vessel Failure (TVF) | 5 years
  cardiac death, MI, clinically indicated TLR
Scaffold Thrombosis | through 5 years
  ARC defined

OTHER OUTCOMES:
Acute success - Procedure success | 7 days
  Acute Success is classified according to the following definitions:
  Procedure success - Successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of < 50% by QCA (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of ischemia driven major adverse cardiac event (MACE) during the hospital stay with a maximum of first seven days post index procedure.
Acute success - Device success | 7 days
  Acute Success is classified according to the following definitions:
  Device success - Successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis < 50% by QCA (by visual estimation if QCA is unavailable). Standard pre-dilation catheters and post-dilatation catheters (if applicable) may be used. Bailout subjects will be included as device success only if the above criteria for clinical device success are met.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Abizaid, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Stefan Verheye, MD, PhD, Principal Investigator — AZ Middelheim Hospital; John Ormiston, MD, Principal Investigator — Auckland City Hospital; Joachim Schofer, MD, PhD, Principal Investigator — Universitäres Herz- und Gefäßzentrum
Locations (13):
- Belgium (2):
  - AZ Middelheim Hospital, Antwerp
  - St. - Jan Ziekenhuis Z.O.L., Genk
- Brazil (2):
  - Instituto Dante Pazzanese, São Paulo
  - ICT / Instituto Do Coracao Do Triangulo Mineiro, Uberlândia
- Aarhus University Hospital, Skejby, Aarhus N, Denmark
- Germany (2):
  - Charite - Campus Benjamin Franklin, Berlin
  - Universitäres Herz- und Gefäßzentrum, Hamburg
- New Zealand (3):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Mercy Angiography Unit, Auckland
- Poland (3):
  - Polsko-Amerykańskie Kliniki Serca, Dąbrowa Górnicza
  - Centrum Interwencyjnego Leczenia Chorób Serca, Krakow
  - Jagiellonian University, Krakow

REFERENCES:
- [Derived] Abizaid A, Costa RA, Schofer J, Ormiston J, Maeng M, Witzenbichler B, Botelho RV, Costa JR Jr, Chamie D, Abizaid AS, Castro JP, Morrison L, Toyloy S, Bhat V, Yan J, Verheye S. Serial Multimodality Imaging and 2-Year Clinical Outcomes of the Novel DESolve Novolimus-Eluting Bioresorbable Coronary Scaffold System for the Treatment of Single De Novo Coronary Lesions. JACC Cardiovasc Interv. 2016 Mar 28;9(6):565-74. doi: 10.1016/j.jcin.2015.12.004. PMID 27013155